CLINICAL TRIAL: NCT01117961
Title: Promoting Healthy Weight Gain During Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: California Polytechnic State University-San Luis Obispo (Other); Women and Infants Hospital of Rhode Island (Other); University of California, Berkeley (Other)
Responsible Party: Principal Investigator, Rena R. Wing, Principal Investigator, The Miriam Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: CMTT# 2035-06
Record Dates: First submitted 2010-04-15; First posted 2010-05-06 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Weight Gain
Keywords: Excessive gestational weight gain
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (No Intervention)
- Intervention (Experimental): Lifestyle intervention delivered during pregnancy
  Interventions: Behavioral: Lifestyle

INTERVENTIONS:
Behavioral: Lifestyle — Behavioral lifestyle intervention targeting diet and physical activity to reduce excessive gestational weight gain
  Arms: Intervention

SUMMARY:
Study goal is to determine whether behavioral lifestyle intervention during pregnancy can reduce the number of women who exceed the Institute of Medicine recommendations for weight gain during pregnancy.

It is hypothesized that the intervention will reduce the number of women who exceed weight gain guidelines relative to standard care. The investigators also expect the intervention to reduce the proportion of women exceeding weight gain guidelines in both normal weight and overweight groups.

ELIGIBILITY:
Inclusion Criteria:

* non-smoking, adults,
* < 16 weeks gestation

Exclusion Criteria:

* medical comorbidities

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 401 (Actual)
Dates: Start 2007-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Percentage of women above the Institute of Medicine Guidelines for gestational weight gain | 40 weeks
  Objective measures of weight collected by trained staff on calibrated scales at study entry and after delivery to classify women as above or below the Institute of Medicine Guidelines for gestational weight gain

SECONDARY OUTCOMES:
Behavioral measures | 40 weeks
  The Block Food Frequency questionnaire and Paffenbarger physical activity questionnaire will be used to assess diet and exercise behavior.

REFERENCES:
- [Derived] Mercado A, Marquez B, Abrams B, Phipps MG, Wing RR, Phelan S. Where Do Women Get Advice About Weight, Eating, and Physical Activity During Pregnancy? J Womens Health (Larchmt). 2017 Sep;26(9):951-956. doi: 10.1089/jwh.2016.6078. Epub 2017 May 19. PMID 28525293
- [Derived] Phelan S, Phipps MG, Abrams B, Darroch F, Grantham K, Schaffner A, Wing RR. Does behavioral intervention in pregnancy reduce postpartum weight retention? Twelve-month outcomes of the Fit for Delivery randomized trial. Am J Clin Nutr. 2014 Feb;99(2):302-11. doi: 10.3945/ajcn.113.070151. Epub 2013 Nov 27. PMID 24284438
- [Derived] Phelan S, Phipps MG, Abrams B, Darroch F, Schaffner A, Wing RR. Randomized trial of a behavioral intervention to prevent excessive gestational weight gain: the Fit for Delivery Study. Am J Clin Nutr. 2011 Apr;93(4):772-9. doi: 10.3945/ajcn.110.005306. Epub 2011 Feb 10. PMID 21310836